CLINICAL TRIAL: NCT06600607
Title: A Randomized, Double-Blind, Placebo-Controlled Crossover Study to Evaluate the Pharmacodynamic Effects of Pregabalin in Healthy Male Adults
Brief Title: Pharmacodynamic Study of 300mg Pregabalin vs Placebo in Healthy Male Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Latigo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LTG-OBS-102
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Pain Detection; Pain Threshold
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Schedule A (Other): participants receive pregabalin 300mg in treatment period 1, and receive placebo in treatment period 2
  Interventions: Drug: pregabalin 300 mg; Other: Placebo
- Schedule B (Other): participants receive placebo in treatment period 1, and receive pregabalin 300mg in treatment period 2
  Interventions: Drug: pregabalin 300 mg; Other: Placebo

INTERVENTIONS:
Drug: pregabalin 300 mg — pregabalin is an FDA-approved anticonvulsant medication commonly used to treat nerve pain
Other: Placebo — biologically inactive placebo comparator

SUMMARY:
This is a randomized, double-blind, placebo-controlled within-participant crossover study in healthy male participants 18-55 years of age to assess pain tolerance during a cold pressor test.

The study will be conducted at a single center in New Zealand.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants aged 18 to 55 years, inclusive, at the time of signing the informed consent.
2. Overtly healthy with no clinically relevant abnormalities based on the medical history, physical examinations, clinical laboratory evaluations, and 12-lead ECG that, in the opinion of the investigator, would affect participant safety.
3. Body mass index (BMI) within the range of 18-32 kg/m2 (inclusive).
4. Male participants are eligible to participate if they agree to refrain from donating semen. Plus, agree to use a male condom when having sexual intercourse with woman of childbearing potential or women who are currently pregnant.
5. Capable of giving signed informed consent.

Exclusion Criteria:

1. Inability to take oral medications or gastrointestinal abnormalities potentially impacting absorption.
2. Clinically significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the investigator, unacceptably increase the participant's risk by participating in the study.
3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST), >1.5 x upper limit of normal (ULN) at Screening.
4. Total bilirubin > 1.5 x ULN (for participants with known Gilbert's syndrome these criteria only apply if total bilirubin > 1.5 x ULN as long as direct bilirubin is ≤ 1.5 x ULN) at Screening.
5. Estimated glomerular filtration rate (eGFR) <80 mL/min based on serum creatinine levels using the 2021 chronic kidney disease epidemiology (CKD-EPI) creatinine equation at Screening.
6. Creatinine phosphokinase is ≤ 2 × ULN at Screening.
7. Any of the protocol defined abnormalities on 12-lead ECG or blood pressure (BP) at Screening, confirmed by repeat.
8. Use of prescription drugs ≤ 14 days (or 5 half-lives of the drug, whichever is longer) prior to Day 1, use of over-the-counter drugs, herbal medications, or vitamin supplements ≤ 7 days (or 5 half-lives of the drug, whichever is longer) prior to Day 1 or use of antibiotics and systemic steroids ≤ 28 days prior Day 1. The Sponsor may allow exceptions only if the medication's administration is deemed unlikely to confound safety.
9. Any vaccination ≤ 14 days prior to Day 1 or anticipated vaccination while participating in the study.
10. Receipt of an investigational product or device, or participation in a drug research study ≤ 28 days (or 5 half-lives of the drug, whichever is longer) prior to Day 1.
11. Receipt of an investigational biologic / monoclonal antibody within 180 days (or 5 half-lives, whichever is longer) prior to Day 1.
12. Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) at Screening.
13. Presence of positive hepatitis C antibody test result at Screening.
14. Positive for Coronavirus Disease 2019 (COVID-19) suggesting active infection at Screening or on Day 1.
15. Positive human immunodeficiency virus (HIV) at Screening.
16. Presence of any condition for which pregabalin administration is contraindicated.
17. Smoking, vaping or use of tobacco or any products containing nicotine ≤ 14 days prior to Day 1.
18. Consumption of alcohol within 48 hours prior to Day 1 and/or food and beverages containing methylxanthines (caffeinated coffee, caffeinated tea, caffeinated soda, and chocolate) within 48 hours of Day 1, and grapefruit, grapefruit juice, Seville oranges, or Seville orange juice ≤ 14 days prior to Day 1.
19. Positive urine drug screen, urine cotinine test, or alcohol breath test at Screening or on Day 1.
20. Donation of over 500 mL blood ≤ 3 months prior to Day 1.
21. Has known psychiatric disorders that would interfere with the cooperation with the requirements of the study.
22. Participant is under legal custodianship.
23. Pain conditions that may require analgesic treatment during the study period/history of opioid medication use.
24. Hand/arm/skin conditions impacting ability to participate in cold pressor assessment.
25. Recent serious injury, surgical procedure, or medical condition which, in the opinion of the investigator, unacceptably increases the participant's risk by being included in the study.
26. Meets protocol defined Pain Tolerance Threshold (PTT) in any of the 5 predose cold pressor tests.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline pain score after dosing with pregabalin vs. placebo | 0-12 hours during each treatment period
  Numerical Pain Rating Scale (NPRS) will be assessed during Cold Pressor Tests at various time points for time to reach Pain Detection Threshold (PDT) and time to reach Pain Tolerance Threshold (PTT)
Time to reach Pain Detection Threshold (PDT) and Pain Tolerance Threshold (PTT) after dosing with pregabalin vs placebo | 0-12 hours during each treatment period
  Stopwatches will be used during each cold pressor test to determine time for subject to reach PDT and PTT

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No